CLINICAL TRIAL: NCT06123169
Title: Postoperative Anti-infective Strategy Following Pancreaticoduodenectomy in Patients With Preoperative Biliary Stent
Acronym: FRENCH24 ANIS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/0423/HP; 2021-006991-18 (EudraCT Number)
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pancreaticoduodenectomy; Antibiotherapy
MeSH Terms: interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broad spectrum antibioprophylaxis (Active Comparator): Antibioprophylaxis with Piperacillin-tazobactam during DPC.
  Interventions: Drug: Antibioprophylaxis (Piperacillin-tazobactam)
- Broad spectrum antibiotherapy (Experimental): 5 days Antibiotherapy (Piperacillin-tazobactam) from surgery.
  Interventions: Drug: 5 days Antibiotherapy (Piperacillin-tazobactam)

INTERVENTIONS:
Drug: Antibioprophylaxis (Piperacillin-tazobactam) — antibiotic prophylaxis during surgery
  Other Names: Control arm
  Arms: Broad spectrum antibioprophylaxis
Drug: 5 days Antibiotherapy (Piperacillin-tazobactam) — 5 days Antibiotherapy from surgery
  Other Names: experimental arm
  Arms: Broad spectrum antibiotherapy

SUMMARY:
The main objective of the study is to compare 2 broad-spectrum antibiotic (Piperacillin / Tazobactam) treatment modalities, following pancreaticoduodenectomy in patients with preoperative biliary stent, to demonstrate the superiority of a 5-day post-operative antibiotic therapy to antibiotic prophylaxis on the occurrence of surgical site infections (SSI)

DETAILED DESCRIPTION:
Despite cumulative efforts in surgery and perioperative management, the morbi-mortality rates of pancreatoduodenectomy (PD) remain high. The most frequent complications were sepsis and infectious complications 44%, hemorrhagic complications 36.6%, pulmonary complications 35.2%, shock 29.8% and pancreatic fistula 27.9%.

PD is a technically complex procedure with substantial associated morbidity and mortality. Infectious complications have been reported to occur in as many as 30% of patients following open PD.

Biliary colonization that arises from preoperative procedures for biliary drainage closely predicts infectious complications following PD. Besides biliary intervention, nutritional reserve and biliary or pancreatic anastomotic leaks are common factors linked to developing infectious complications following PD.

D'Angelica et al. Recently demonstrated the superiority of Piperacillin-tazobactam compared with cefoxitin as antimicrobial prophylaxis for PD: a randomized clinical trial in JAMA, with a significant reduction of postoperative SSI rate.

One of the main risk factors for infectious complications and especially surgical site infections, but also post-operative pancreatic fistula is bacteriobilia, defined by the bile contamination by microorganism(s) related to preoperative biliary drainage.

A significant decrease in all-type SSI and organ-space SSI with Broad spectrum antibiotics was observed after open PD, as reported by Kone et al. or De Grandi et al. According to Kone et al. on subgroup analysis, only patients with preoperative biliary stents and/ or jaundice (61% of PD patients) had an association between Broad-abx and decreased SSI. Numbered of surgeons modified their antibiotic usage in this setting of preoperative biliary drainage, as we also observed in France, where more than 50% prescribed a broad spectrum antibiotherapy intraoperatively only (antibioprophylaxis) or for 3 to 5 days.

The aim of this study is to determine whether a prophylactic treatment used only during surgery, or for 5 days with this treatment, in the clinical context of PD after biliary drainage, is effective in reducing surgical complications, particularly infectious ones.

Such results could reduce the need for prolonged anti-infectious treatments and reoperations (surgical and radiological). Hospital stays could also be shortened, with a positive impact on your quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Planned pancreaticoduodenectomy for periampullary neoplasms
* Endoscopic or radiological pre-operative biliary drainage
* Age ≥ 18 years old
* Patient able to comply with the study protocol, in the investigator's judgment
* Patient affiliated with, or beneficiary of a social security (national health insurance) category
* Person of full age having read and understood the information letter and signed the consent form
* Women of childbearing potential (a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile) with hightly effective contraception (Cf. CTFG) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system ( IUS), bilateral tubal occlusion, vasectomised partner, sexual abstinence) since 1 month and during the duration of the study and a negative blood pregnancy test by beta-HCG at inclusion.
* Women permanently sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
* Postmenopausal women: A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Exclusion Criteria:

* Contraindication to PIPERACILLIN/TAZOBACTAM PANPHARMA 4g / 500mg powder for solution for injection in accordance with its SmPC
* Patients allergic to beta-lactam antibiotics
* Others pancreatic resection
* Absence of preoperative biliary drainage
* Surgical or anaesthesiological contra-indications:
* non-controlled congestive heart failure - non-treated angina - recent myocardial infarction (in the previous year) - non-controlled AHT (SBP >160 mm or DBP > 100 mm, despite optimal drug treatment), long QT
* major non-controlled infection
* severe liver failure
* Medical, geographical, sociological, psychological or legal conditions that would not permit the patient to complete the study or sign informed consent
* Any significant disease, which, in the investigator's opinion, would exclude the patient from the study
* Pregnant or parturient or breastfeeding woman or absence of contraceptionn
* Person deprived of liberty by administrative or judicial decision or person placed under judicial protection, under guardianship or supervision
* Simultaneous participation in another interventional research with the same primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
presence of an organ/space SSI | 90 days after the surgery
  The primary End Point is the presence of an organ/space SSI determined according to the Centers for Disease Control and Prevention's national nosocomial infections surveillance system. Organ/space SSIs include postoperative pancreatic fistula (POPF) and bile leakage, with positive culture results.

SECONDARY OUTCOMES:
Infectious complications at post-operative | day 90
  Overall postsurgical morbidity, graded according to the Dindo/Clavien classification and CCI score
Correlation between post-operative bacteriological samples and intraoperative bile samples | day 90
  Correlation between post-operative bacteriological samples and intraoperative bile samples (presence of bacterial strains)
Bacteriological resistance profiles | day 90
  Incidence of fungal contamination
Correlation between bacteriological and fungal contaminations | day 90
  Correlation between bacteriological and fungal contaminations (presence of bacterial strains and fungal contamination)
Specific morbidity due to pancreatic fistula, graded according to the International Study Group of Pancreatic Fistula (ISGPF) criteria | day 90
  Specific morbidity due to pancreatic fistula, graded according to the International Study Group of Pancreatic Fistula (ISGPF) criteria
Readmission rates and Duration of hospitalization | day 90
  Readmission rates and Duration of hospitalization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwarz L, Gillibert A, Rondeaux J, Lacroix E, Sa Cunha A, Joannes-Boyau O. Study protocol of the FRENCH24-ANIS study: postoperative anti-infective strategy following pancreaticoduodenectomy in patients with preoperative biliary stents-an intergroup FRENCH-ACHBT-SFAR prospective randomized controlled trial. BMC Surg. 2024 Aug 22;24(1):237. doi: 10.1186/s12893-024-02507-y. PMID 39169298